CLINICAL TRIAL: NCT02068534
Title: A Qualitative and Quantitative Analysis on the Living History of Survivors From Charcoal-burning Suicide
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yi-Ju Pan, visiting doctor, Far Eastern Memorial Hospital
Other Study IDs: 102122-F
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Suicide
Keywords: in-depth individual interview; charcoal-burning suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- survivors from charcoal-burning suicide: survivors from charcoal-burning suicide and at least above 20 years old.

SUMMARY:
The current study aims to explore the risk factors, protective factors, resilient factors, and factors jeopardizing the recovery progress on survivors from charcoal-burning suicide. To this end, an in-depth individual interview and Mini-Mental State Examination(MMSE) will be used to acquire the first-hand information on the attempters. As well, a more comprehensive neuropsychological test, WAIS III, will be administered at 3-month, 6-month, and 12-month after the index suicide attempt.

ELIGIBILITY:
Inclusion Criteria:

* above 20 years old, survivors from charcoal-burning suicide.

Exclusion Criteria:

* under 20 years old
* survivors from other kind of suicide
* prisoner
* suffer from a serious illness
* foreigner/ can't speak Chinese
* the people who can't express themselves
* can not be interviewed in FEMH
* people with severe physical or psychological symptoms

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: survivors from charcoal-burning suicide
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
MMSE score | once

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ju Pan, Ph. D., Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei City, Taiwan